CLINICAL TRIAL: NCT04162028
Title: Pre-hospital Utilization of Nebulized Sub-dissociative Dose Ketamine for Managing Acute Traumatic Extremity Pain: a Prospective Observational Study
Brief Title: Pre-hospital Nebulized Ketamine for Pain
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigators not interested any more in the study
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-10-08
Record Dates: First submitted 2019-11-04; First posted 2019-11-13 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nebulized Ketamine (Experimental): sub-dissociative dose ketamine administered prehospitally via breath-actuated nebulizer at 1.0 mg/kg for patients with acute pain
  Interventions: Drug: Nebutlized Ketamine

INTERVENTIONS:
Drug: Nebutlized Ketamine — The PK-BAN package will be opened and weight -based dose of ketamine will be administered to the patient via BAN. The medication will be delivered with a minimum time of 5 min and maximum time of 15 min.
  Other Names: ketamine

SUMMARY:
In the situation when intravenous access is not readily available or unobtainable, or when prehospital delays to obtain intravenous access are not warranted, sub-dissociative dose ketamine can be administered via intranasal (IN) route. The data supporting IN is not set on the optimum intranasal dose (range 0.75-1 mg/kg) and frequencies of administration. In addition, IN administration of SDK for adult patients in the ED requires a highly concentrated solution that is not routinely stock in the ED. Hence, another non-invasive route exists such as nebulization via a Breath-Actuated Nebulizer which allows a controlled patient-initiated delivery of analgesics in titratable fashion.

Nebulized administration of ketamine however, has only been studied in the areas of acute postoperative pain management, cancer palliation, and status asthmaticus therapy (ref). To our knowledge, there are no prospective randomized trials that evaluated a role of nebulized SDK role in managing acute pain due to extremity trauma in the prehospital arena.

We aim to evaluate analgesic efficacy and safety of sub-dissociative dose ketamine administered prehospital via breath-actuated nebulizer at 1.0 mg/kg for patients with acute traumatic extremity injuries.

DETAILED DESCRIPTION:
Ketamine is a non-competitive N-methyl-D-aspartate (NMDA)/glutamate receptor complex antagonist that decreases pain by diminishing central sensitization, hyperalgesia, and "wind-up" phenomenon at the level of the spinal cord (dorsal ganglion) and central nervous system Ketamine administration in sub-dissociative doses (0.1-0.3 mg/kg) in prehospital settings and in the ED results in effective pain relief in patients with acute traumatic and non-traumatic pain, chronic non-cancer and cancer pain, and in patients with opioid-tolerant pain by virtue of providing anti-hyperalgesia, anti-allodynia, and anti-tolerance. Two commonly employed strategies of SDK administration in the ED include an intravenous push (IVP) dose (over 2-5 minutes), which is associated with relatively high rates of minor but bothersome psycho-perceptual side effects (feeling of unreality and dizziness), or short infusion (SI) given over 15 minutes with significantly reduced rates of unreality and preserved analgesic efficacy.

In the current study the investigators hypothesize that sub-dissociative-dose ketamine administered as a single agent via breath actuated nebulizer at the dose of 1.0 mg/kg will provide significant pain relief with minimal rates of side effects for patients with acute traumatic extremity injuries and will allow for alternative administration of effective analgesia especially in those settings for which intravenous or intraosseous routes are difficult or not necessary or when a delay in patient transport to a hospital is not ideal.

The primary outcome of this trial is the percent reduction in participant's pain scores at 30 minutes post medication administration.

STUDY DESIGN

Subjects: Patients 18 years of age and older transported by prehospital care providers to the ED with acute traumatic extremity injuries with a pain score of 5 or more on a standard 11- point (0 to 10) numeric rating scale. Patients will be enrolled by Emergency Medical Services (EMS) providers of Maimonides Medical Center (MMC) who are operating under the New York City 9-1-1 Regional Emergency Medical Advisory Committee (REMAC) auspices. Patient screening, enrollment, and data collection will be performed initially by advanced life support (ALS) paramedics and subsequently completed by study investigators upon arrival to the MMC emergency department. Emergency department pharmacist investigators will prepare PK-BAN packages that will be assigned to every ALS ambulance at the start of shift. The package will include a single ketamine 50mg/ml vial, blunt-tip needle and syringe, BAN device/tubing, and data collection sheet.

Eligibility Criteria: Patients 18 years of age and older with acute traumatic extremities injuries with a score of 5 or more on a standard 11- point (0 to 10) numeric rating scale.

Exclusion criteria will include altered mental status, allergy to ketamine, pregnant patients, weight greater than 150 kg, unstable vital signs (systolic blood pressure <90 or>180 mm Hg, pulse rate <50 or >150 beats/min, and respiration rate <10 or >30 breaths/min), and past medical history of alcohol or drug abuse, or schizophrenia.

Design: This is a prospective, observational study evaluating analgesic efficacy and safety of sub-dissociative dose ketamine of 1.0 mg/kg administered via breath-actuated nebulizer

Data Collection Procedures: Each patient will be approached by advanced life support (ALS) paramedics for acquisition of written informed consent and Health Insurance Portability and Accountability Act authorization after meeting study eligibility criteria. In case of severe pain (extremis), a verbal consent will suffice the initial administration of the SDK with subsequent signing of the informed consent upon arrival to the ED. Baseline pain score will be determined with an 11-point numeric rating scale (0 to 10), described to the patient as "no pain" being 0 and "the worst pain imaginable" being 10. An ALS paramedic will record the patient's body weight and baseline vital signs. The PK-BAN package will be opened and weight -based dose of ketamine will be administered to the patient via BAN. The medication will be delivered with a minimum time of 5 min and maximum time of 15 min. An ALS Paramedic record pain scores, vital signs, and adverse effects at 15 and 30 minutes. If patients reported a pain numeric rating scale score of 5 or greater and requested additional pain relief, a second (equivalent to the first dose) of SDK via BAN will be administered to the patient in a blinded fashion. In situations when nebulized SDK will fail to achieve acceptable (by patient) pain relief or patient will refuse to continue nebulized SDK treatment, morphine at 0.1 mg/kg IV/IO/IM (not to exceed 5mg) will be administered as a rescue analgesic with an option for one repeat dose (maximum total dose is 10mg).

All data will be recorded on data collection sheets, including patients' sex, demographics, medical history, and vital signs and entered into SPSS (version 24.0; IBM Corp) by the research manager. Confirmation of written consent acquisition for all participants and statistical analyses will be conducted by the research manager and statistician, who would work independent of any data collection.

Patients will be closely monitored for any change in vital signs and for adverse effects during the entire study period (up to 2 hours) by study investigators after arrival to the ED. Common adverse effects that are associated with sub-dissociative dose ketamine are feeling of unreality, dizziness, nausea, vomiting, and sedation.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and older
* acute traumatic extremities injuries
* a score of 5 or more on a standard 11- point (0 to 10) numeric rating scale.

Exclusion Criteria:

* Patients with altered mental status,
* allergy to ketamine, pregnant patients,
* weight greater than 100 kg,
* unstable vital signs (systolic blood pressure <90 or>180 mm Hg,
* pulse rate <50 or >150 beats/min,
* respiration rate <10 or >30 breaths/min),
* inability to consent,
* past medical history of alcohol or drug abuse
* schizophrenia.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Change in Pain Scores | 30 minutes
  The primary outcome will include a percentage of patients achieving a 20% or greater change in pain scores on numeric rating pain scale (NRS) ranging form 0 no pain to 20 severe pain for the baseline to 30 minutes post-analgesic administration.

SECONDARY OUTCOMES:
Rescue Analgesia | 30 minutes
  The secondary outcomes will include a need for second or third dose, a need for rescue analgesia at either 15 and 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT04162028/Prot_SAP_000.pdf